CLINICAL TRIAL: NCT03983941
Title: Comparison of Postoperative Analgesic Efficacy of Adductor Canal Block With IPACK Versus Adductor Canal and Popliteal Sciatic Nerve Block in Patients Undergoing Arthroscopic Anterior Cruciate Ligament Reconstruction
Brief Title: IPACK Versus Popliteal Sciatic Nerve Block in ACL Reconstruction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI leaving the institution, no subjects enrolled since 2019, and no other PI interested in taking it over.
Sponsor: Sujana Dontukurthy (Other)
Responsible Party: Sponsor-Investigator, Sujana Dontukurthy, Clinical Assistant Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000281
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Anterior Cruciate Ligament Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- FNB-AC + Sciatic nerve block (Active Comparator): Patients will receive up to 20 mL of 0.2% ropivacaine for FNB-AC and up to 20 mL of 0.2% ropivacaine for sciatic nerve block under ultrasound guidance.
  Interventions: Drug: Ropivacaine injection
- FNB-AC + IPACK (Experimental): Patients will receive up to 20 mL of 0.2% ropivacaine for FNB-AC and up to 20 mL of 0.2% ropivacaine for posterior knee capsular infiltration under ultrasound guidance (IPACK)
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: Ropivacaine injection — Total dose not to exceed 3 mg/kg of ropivacaine.

SUMMARY:
This is a prospective study comparing femoral nerve block plus sciatic nerve block to femoral nerve block plus infiltration of the posterior knee capsule (IPACK) in patients undergoing arthroscopic anterior cruciate ligament reconstruction. Femoral nerve block via the adductor canal (FNB-AC) with IPACK may provide effective analgesia while avoiding the motor block involved with sciatic nerve block. The lack of motor block is important to facilitate postoperative ambulation and physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 21 years of age
* American Society of Anesthesiologists physical status I and II
* Undergoing elective anterior cruciate ligament reconstruction

Exclusion Criteria:

* They are unable or unwilling to take part in the study
* History of allergy to any of the medications administered for the nerve block
* Contraindication to peripheral nerve block
* Patients who are unable to understand instructions or questions related to the study or the families required language interpretation
* Patients who consume opioid medications for more than three days per week for more than a month prior to surgery

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FNB-AC + Sciatic Nerve Block | FNB-AC + IPACK
Started | 2 | 5
Completed | 2 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FNB-AC + Sciatic Nerve Block | FNB-AC + IPACK | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 3 | 5
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 15.8 [14.6 to 16.9] | 17 [14 to 20.8] | 16.7 [14 to 20.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Average Post-operative Pain Score
Description: Visual Analogue Scale (VAS) pain scores (0 being no pain and 10 being worst pain) from arrival to post-anesthesia care unit (PACU) to 48 hours after discharge from surgery center.
Time Frame: Immediately post-operatively and up to 48 hours post-discharge, an average of 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FNB-AC + Sciatic Nerve Block | FNB-AC + IPACK
Number analyzed (Participants) | 2 | 5
score on a scale | 4.7 (3.368) | 4 (2.905)

2. Secondary Outcome: Number of Opioid Doses Administered
Description: Number of doses of narcotic pain medicine administered during surgery and up to 48 hours after discharge from surgery center.
Time Frame: Intra-operative and up to 48 hours post-discharge, an average of 48 hours
Measure: Mean (Full Range); unit: opiod doses administered
Arm/Group | FNB-AC + Sciatic Nerve Block | FNB-AC + IPACK
Number analyzed (Participants) | 2 | 5
opiod doses administered | 5.5 [4 to 7] | 3.8 [2 to 5]

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | FNB-AC + Sciatic Nerve Block | FNB-AC + IPACK
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 0/2 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT03983941/Prot_SAP_000.pdf